CLINICAL TRIAL: NCT03639610
Title: A Study of the Pharmacokinetics of Melphalan During Treatment With Melflufen and Dexamethasone in Patients With Relapsed Refractory Multiple Myeloma and Impaired Renal Function
Brief Title: PK of Melphalan During Treatment With Melflufen and Dexamethasone in Patients With RRMM and Impaired Renal Function
Acronym: BRIDGE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to terminate the study following an FDA request of a partial clinical hold.
Sponsor: Oncopeptides AB (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP-107; 2018-000478-31 (EudraCT Number)
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Renal Impairment; Multiple Myeloma
MeSH Terms: conditions — Renal Insufficiency; Multiple Myeloma | interventions — melflufen; L-melphalanyl-p-L-fluorophenylalanine ethyl ester; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Arms differed based on patients' level of renal function (moderate or severe impairment) and starting dose of melflufen.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1a (Experimental): Patients with moderate renal impairment (eGFR ≥30 to <45 mL/min/1.73m²) and a starting dose of melflufen of 40 mg
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Cohort 1b (Experimental): Patients with moderate renal impairment (eGFR ≥30 to <45 mL/min/1.73m²) and a starting dose of melflufen of 30 mg
  Interventions: Drug: Melflufen; Drug: Dexamethasone
- Cohort 2a (Experimental): Patients with severe renal impairment (eGFR ≥15 to <30 mL/min/1.73m²) and a starting dose of melflufen of 20 mg
  Interventions: Drug: Melflufen; Drug: Dexamethasone

INTERVENTIONS:
Drug: Melflufen — Melflufen was distributed in the European Union (EU) as a powder for concentrate for solution for infusion; in the US, it was distributed as a powder for injection. Melflufen was administered as a 30-minute intravenous infusion on Day 1 of every 28-day cycle via a central catheter.
  Other Names: Melphalan flufenamide
Drug: Dexamethasone — Tablets. Administered orally on Days 1, 8, 15, and 22 of each 28-day cycle. Dose of 40 mg for patients aged <75 years. Dose of 20 mg for patients aged ≥75 years.

SUMMARY:
This was a multicenter study of the pharmacokinetics (PK) of melphalan during treatment with melflufen and dexamethasone in patients with relapsed refractory multiple myeloma (RRMM) and impaired renal function.

DETAILED DESCRIPTION:
This was a multicenter study assessing the safety, tolerability, and efficacy of melflufen given on Day 1 of a 28-day cycle, together with weekly dexamethasone, in patients with relapsed multiple myeloma or RRMM and impaired renal function, as well as the relationship between renal function and PK parameters for the active metabolite melphalan.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 years or older, at the time of signing the informed consent;
2. A prior diagnosis of multiple myeloma (MM) with documented disease progression in need of treatment at time of screening;
3. Received at least 2 prior lines of therapy;
4. Measurable disease defined as any of the following:

   * Serum monoclonal protein ≥0.5 g/dL by serum protein electrophoresis (SPEP).
   * ≥200 mg/24 hours of monoclonal protein in the urine on 24-hour urine electrophoresis (UPEP)
   * Serum free light chain (SFLC) ≥10 mg/dL AND abnormal serum kappa to lambda free light chain ratio
5. Life expectancy of ≥6 months;
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤2. (Patients with lower performance status based solely on bone pain secondary to MM may be eligible following consultation and approval of the medical monitor);
7. Patient is a female of childbearing potential (FCBP)* with a negative serum or urine pregnancy test prior to initiation of therapy and agrees to practice appropriate methods of birth control, or the patient is male and agrees to practice appropriate methods of birth control;
8. Ability to understand the purpose and risks of the study and provide signed and dated informed consent;
9. 12-lead electrocardiogram (ECG) with QT interval calculated by Fridericia Formula (QTcF) interval of ≤470 msec;
10. Renal function: Estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula on 2 consecutive screening evaluations. Patients meeting criteria for Screening 1, must also meet criteria for Screening 2 following optimal hydration (as determined by the investigator). Screening 2 must be on or as close as possible to treatment start date (preferably <24-48 hours) but cannot exceed 72 hours.

    • Cohort 1 (a and b): Screening 1: eGFR between ≥25 mL/min/1.73m² to <45 mL/min/1.73m². Screening 2: eGFR between ≥30 mL/min/1.73m² to <45 mL/min/1.73m².

    • Cohort 2 (a and b): Screening 1: eGFR between ≥10 mL/min/1.73m² to <35 mL/min/1.73m². Screening 2: eGFR between ≥15 mL/min/1.73m² to <30 mL/min/1.73m².

    Cohort 2b will only be enrolled following approval of Data Safety Monitoring Committee (DSMC) after evaluating data from Cohort 1a, 1b and 2a.

    Patients with fluctuating values of eGFR may be eligible following consideration of additional assessments in consultation with the medical monitor.
11. The following laboratory results must be met during screening (within 21 days) and immediately before study drug administration on Cycle 1 Day 1:

    * Absolute neutrophil count (ANC) ≥1,000 cells/mm³ (1.0 x 10⁹/L) (Growth factors cannot be used within 10 days [14 days for pegfilgrastim] prior to initiation of therapy)
    * Platelet count ≥75,000 cells/mm³ (75 x 10⁹/L) (without required transfusions during the 10 days prior to initiation of therapy)
    * Hemoglobin ≥8.0 g/dL (red blood cell [RBC] transfusions are permitted)
    * Total Bilirubin ≤1.5 x upper limit of normal (ULN), or higher in patients diagnosed with Gilbert's syndrome, that have been reviewed and approved by the medical monitor
    * Aspartate transaminase / serum glutamic oxaloacetic transaminase (AST / SGOT) and alanine transaminase / serum glutamic pyruvic transaminase (ALT / SGPT) ≤3.0 x ULN;
12. Must have, or be willing to have, an acceptable central catheter. (Port a cath, peripherally inserted central catheter [PICC] line, or central venous catheter).

Footnote

*FCBP is any sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal (not having menstrual cycles due to cancer therapy does not rule out childbearing potential) for at least 24 consecutive months.

Exclusion Criteria:

1. Primary refractory disease (i.e., never responded with ≥ minimal response [MR] to any prior therapy);
2. Evidence of mucosal or internal bleeding and/or platelet transfusion refractory (platelet count fails to increase by >10,000 cells/mm³ [10.0 x 10⁹/L] after a transfusion of an appropriate dose of platelets);
3. Any medical conditions that, in the Investigator's opinion, would impose excessive risk to the patient or would adversely affect his/her participating in this study. Examples of such conditions are: a significant history of cardiovascular disease (e.g., myocardial infarction, significant conduction system abnormalities, uncontrolled hypertension, ≥Grade 3 thromboembolic event in the last 6 months);
4. Known active infection requiring parenteral or oral anti-infective treatment within 14 days of initiation of therapy;
5. Other malignancy diagnosed or requiring treatment within the past 3 years with the exception of adequately treated basal cell carcinoma, squamous cell skin cancer, carcinoma in-situ of the cervix or breast or very low and low risk prostate cancer in active surveillance;
6. Pregnant or breast-feeding females;
7. Serious psychiatric illness, active alcoholism, or drug addiction that may hinder or confuse compliance or follow-up evaluation;
8. Known human immunodeficiency virus or active hepatitis B or C viral infection;
9. Concurrent symptomatic amyloidosis or plasma cell leukemia;
10. POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes);
11. Previous cytotoxic therapies, including cytotoxic investigational agents, for MM within 3 weeks (6 weeks for nitrosoureas) prior to initiation of therapy. The use of live vaccines within 30 days before initiation of therapy. Immunomodulatory drugs (IMiDs), proteasome inhibitors (PIs) or corticosteroids within 2 weeks prior to initiation of therapy. Other investigational therapies and monoclonal antibodies (mAb) within 4 weeks of initiation of therapy. Prednisone up to but no more than 10 mg orally once daily (q.d.) or its equivalent for symptom management of comorbid conditions is permitted but dose should be stable for at least 7 days prior to initiation of therapy;
12. Residual side effects to previous therapy >Grade 1 prior to initiation of therapy (Alopecia any grade and/or neuropathy Grade 2 without pain are permitted);
13. Prior peripheral stem cell transplant within 12 weeks of initiation of therapy;
14. Prior allogeneic stem cell transplantation with active graft-versus-host-disease;
15. Prior major surgical procedure or radiation therapy within 4 weeks of initiation of study therapy (this does not include limited course of radiation used for management of bone pain to be completed within 7 days of initiation of study therapy). Plasmapheresis is not permitted within 14 days of initiation of therapy;
16. Known intolerance to steroid therapy;
17. Prior renal transplant;
18. Currently in need of renal dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- Czechia (3):
  - University Hospital Brno, Clinic of Internal Medicine - Hematology and Oncology, Brno
  - University Hospital Olomouc, Clinic of Hemato-Oncology, Olomouc
  - General University Hospital in Prague, 1st Internal Clinic - Clinic of Hematology, Prague
- Greece (3):
  - General Hospital of Athens "Evangelismos", Athens
  - General Hospital of Athens Alexandra, Therapeutic Clinic, Athens
  - University General Hospital of Patras, Pátrai
- Poland (4):
  - Nasz Lekarz Medical Outpatient Clinics Slawomir Jeka, Torun, Torun
  - Maria Sklodowska-Curie Institute of Oncology, Branch in Gliwice, Department of Bone Marrow Transplantation and Hematologic Oncology, Gliwice
  - Independent Public Healthcare Facility Municipal Hospitals, Department of Hematology, Katowice
  - Independent Public Teaching Hospital No.1 in Lublin, Department of Hematooncology, Bone Marrow Transplantation and Chemotherapy, Lublin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient (in Cohort 1a) received their first dose of study drug on 17 September 2018. The last patient (in Cohort 2a) received their first dose of study drug on 29 June 2021.
Pre-assignment Details: All enrolled patients received study treatment and were included in the Safety Analysis Set.
Groups:
- Cohort 1a, Melflufen 40 mg: Patients with moderate renal impairment (eGFR ≥30 to <45 mL/min/1.73m²) and a starting dose of melflufen of 40 mg.
- Cohort 1b, Melflufen 30 mg: Patients with moderate renal impairment (eGFR ≥30 to <45 mL/min/1.73m²) and a starting dose of melflufen of 30 mg.
- Cohort 2a, Melflufen 20 mg: Patients with severe renal impairment (eGFR ≥15 to <30 mL/min/1.73m²) and a starting dose of melflufen of 20 mg.
Period: Overall Study
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Started | 21 | 10 | 4
Completed | 0 | 0 | 0
Not Completed | 21 | 10 | 4
Not completed — Adverse Event | 7 | 1 | 0
Not completed — Physician Decision | 3 | 1 | 0
Not completed — Disease progression | 8 | 5 | 3
Not completed — Study terminated by sponsor | 2 | 1 | 1
Not completed — Patient request to stop treatment | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are shown for the Safety Analysis Set, which is defined as all patients who received at least 1 or partial dose of melflufen or dexamethasone.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg | Total
Number analyzed (Participants) | 21 | 10 | 4 | 35
Age, Continuous [Median (Full Range); unit: years] | 70.0 [52 to 84] | 72.0 [54 to 85] | 62.5 [57 to 76] | 70.0 [52 to 85]
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 4 | 3 | 3 | 10
  ≥65 to ≤75 years | 9 | 5 | 0 | 14
  >75 years | 8 | 2 | 1 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 1 | 16
  Male | 12 | 4 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 10 | 4 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 21 | 10 | 4 | 35
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Greece | 9 | 4 | 3 | 16
  Czechia | 4 | 4 | 1 | 9
  Poland | 8 | 2 | 0 | 10
Baseline height [Median (Full Range); unit: cm] | 165.0 [147 to 181] | 169.0 [155 to 189] | 172.5 [167 to 180] | 168.0 [147 to 189]
Baseline weight [Median (Full Range); unit: kg] | 73.00 [57.3 to 132.0] | 75.25 [54.0 to 140.0] | 85.50 [73.0 to 110.0] | 74.00 [54.0 to 140.0]
Baseline Eastern Cooperative Oncology Group (ECOG) score [Count of Participants; unit: Participants] — ECOG Performance Scale:
  0=Normal activity, fully active, able to carry on all pre-disease performance without restriction. 1=Symptoms, but fully ambulatory, restricted in physically strenuous but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    score = 0 | 11 | 3 | 3 | 17
    score = 1 | 8 | 6 | 1 | 15
    score = 2 | 2 | 1 | 0 | 3
International Staging System (ISS) stage at study entry [Count of Participants; unit: Participants] — ISS Stage Stage I: Serum B2-microglobulin <3.5 mg/L; serum albumin >=3.5 g/dL Stage II: Not ISS Stage I or III. Stage III: Serum B2-microglobulin >=5.5mg/L R-ISS Stage Stage I: ISS Stage I and standard risk chromosomal abnormalities (CA) by interphase by florescent in situ hybridization (iFISH) & normal lactate dehydrogenase (LDH) Stage II: Not R-ISS Stage I or III Stage III: ISS Stage III & either high risk CA by iFISH or high LDH
  Participants
    stage I | 2 | 0 | 0 | 2
    stage II | 9 | 4 | 1 | 14
    stage III | 9 | 6 | 3 | 18
    unknown | 1 | 0 | 0 | 1
Evidence of lytic bone disease at study entry [Count of Participants; unit: Participants]
  Yes | 16 | 9 | 4 | 29
  No | 5 | 1 | 0 | 6
Evidence of extramedullary disease at study entry [Count of Participants; unit: Participants]
  Yes | 1 | 1 | 1 | 3
  No | 20 | 9 | 3 | 32
Disease status at study entry [Count of Participants; unit: Participants]
  Relapsed | 13 | 3 | 2 | 18
  Relapsed-refractory | 8 | 7 | 2 | 17
Time since diagnosis [Median (Full Range); unit: years] | 6.47 [1.1 to 11.1] | 3.82 [0.9 to 8.0] | 5.13 [1.6 to 7.7] | 4.78 [0.9 to 11.1]
Time since most recent relapse/progression [Median (Full Range); unit: months] | 1.12 [0.5 to 9.8] | 1.49 [0.6 to 5.8] | 3.29 [0.9 to 9.3] | 1.25 [0.5 to 9.8]
Baseline estimated glomerular filtration rate (eGFR) [Count of Participants; unit: Participants] — Note that eligibility was based on eGFR measured at Screening, while Baseline measurements are from Cycle 1 Day 1. For some patients, the eGFR value was derived using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula when eGFR was not reported but the corresponding visit serum creatinine value was available.
  Participants
    ≥15 to <30 mL/min/1.73m² | 0 | 2 | 4 | 6
    ≥30 to <45 mL/min/1.73m² | 19 | 8 | 0 | 27
    ≥45 mL/min/1.73m² | 2 | 0 | 0 | 2
Cytogenetics abnormalities by interphase fluorescence in situ hybridization (iFISH) at study entry [Count of Participants; unit: Participants] — The high-risk based on iFISH is defined in case the following abnormalities were found: deletion (17p), gain 1q (+1q), gain (1q21); t (4;14), t(4;14) (p16;q32), t (14;16), t (14;16) (q32;q23), t(14;20), t(14;20) (q32;q11). The standard-risk based on iFISH consists of patients who have a genetic subtype recorded but none of the genetic subtypes categorized as high-risk based on iFISH. The category of unknown consists of patients for whom the iFISH procedure was not done or unevaluable.
  Participants
    High-risk abnormalities | 5 | 5 | 0 | 10
    Standard-risk abnormalities | 16 | 4 | 3 | 23
    Unknown | 0 | 0 | 1 | 1
    Missing | 0 | 1 | 0 | 1
Prior autologous transplant [Count of Participants; unit: Participants] | 9 | 1 | 1 | 11
Number of prior systemic therapy lines [Count of Participants; unit: Participants] — There was one patient who reported 2 prior line of therapies but only one of them was multiple myeloma therapy. However, this exception was not reflected in the database since a minimum of 2 lines were possible to report. Although this patient was enrolled into the study incorrectly, the patient was not excluded from analyses.
  Participants
    2 prior lines of therapy | 5 | 6 | 2 | 13
    3 prior lines of therapy | 7 | 2 | 1 | 10
    4 prior lines of therapy | 9 | 2 | 1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Melphalan
Description: Maximum observed concentration (Cmax)
Time Frame: Samples were drawn 5-10 minutes after the end of infusion, 2-3 hours after the end of infusion, and 5-7 hours after the end of infusion.
Population: Some patients were not evaluable for pharmacokinetics (PK) and were excluded from Cycle 1 and/or Cycle 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
ng/mL
  Cycle 1: number analyzed (Participants) | 13 | 5 | 4
  Cycle 1 | 550.1538 (170.024) | 472.2000 (141.505) | 181.2500 (76.098)
  Cycle 2: number analyzed (Participants) | 9 | 6 | 3
  Cycle 2 | 539.4444 (178.246) | 469.5000 (177.340) | 194.0000 (57.663)

2. Primary Outcome: Tmax of Melphalan
Description: Time of maximum observed concentration (Tmax)
Time Frame: as for outcome 1
Population: Some patients were not evaluable for PK and were excluded from Cycle 1 and/or Cycle 2.
Measure: Median (Full Range); unit: minutes
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
minutes
  Cycle 1: number analyzed (Participants) | 13 | 5 | 4
  Cycle 1 | 38.0000 [35.0000 to 40.0000] | 40.0000 [35.0000 to 45.0000] | 37.0000 [36.0000 to 40.0000]
  Cycle 2: number analyzed (Participants) | 9 | 6 | 3
  Cycle 2 | 37.0000 [35.0000 to 40.0000] | 40.0000 [38.0000 to 40.0000] | 36.0000 [35.0000 to 37.0000]

3. Primary Outcome: Area Under the Curve (0-t) of Melphalan
Description: Area under the concentration-time curve (AUC) from 0h to the last measurable concentration.
Time Frame: as for outcome 1
Population: Some patients were not evaluable for PK and were excluded from Cycle 1 and/or Cycle 2.
Measure: Mean (Standard Deviation); unit: minutes*ng/mL
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
minutes*ng/mL
  Cycle 1: number analyzed (Participants) | 13 | 5 | 4
  Cycle 1 | 78250.3462 (21391.384) | 70303.4400 (16874.787) | 27912.7125 (10385.219)
  Cycle 2: number analyzed (Participants) | 9 | 6 | 3
  Cycle 2 | 74415.5556 (21354.648) | 67458.0000 (19241.040) | 32146.0000 (5804.816)

4. Primary Outcome: Area Under the Curve (Inf) of Melphalan
Description: Area under the concentration-time curve (AUC) from 0 hours to infinity
Time Frame: as for outcome 1
Population: Some patients were not evaluable for PK and were excluded from Cycle 1 and/or Cycle 2.
Measure: Mean (Standard Deviation); unit: minutes*ng/mL
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
minutes*ng/mL
  Cycle 1: number analyzed (Participants) | 13 | 5 | 4
  Cycle 1 | 85123.3635 (22765.646) | 77173.0689 (15347.431) | 31712.9042 (11597.404)
  Cycle 2: number analyzed (Participants) | 9 | 6 | 3
  Cycle 2 | 80365.5468 (22334.049) | 72830.2410 (20632.358) | 39685.8277 (6405.267)

5. Primary Outcome: T1/2 of Melphalan
Description: Elimination half-life of melphalan
Time Frame: as for outcome 1
Population: Some patients were not evaluable for PK and were excluded from Cycle 1 and/or Cycle 2.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
minutes
  Cycle 1: number analyzed (Participants) | 13 | 5 | 4
  Cycle 1 | 89.1390 (15.575) | 98.3568 (27.249) | 109.5502 (22.221)
  Cycle 2: number analyzed (Participants) | 9 | 6 | 3
  Cycle 2 | 87.5544 (15.860) | 90.7844 (14.411) | 136.2193 (13.679)

6. Secondary Outcome: Best Confirmed Response
Description: Best confirmed response required 2 consecutive assessments with the same response result made at any time. In case at the second consecutive assessment (made at any time) the response is higher than the previous one, then confirmed response (linked to the first assessment visit) will be the first one (e.g., PR - VGPR consecutive pair will lead to a PR confirmed response at the first visit). In case the second consecutive response is lower than the first one, then confirmed response (linked to the first assessment visit) will be the second one (e.g. CR-VGPR consecutive pair will lead to a VGPR confirmed response at the first visit).
Time Frame: Patients were assessed for response after each cycle. After discontinuation of therapy, patients continued to be assessed until documented progression (confirmed on 2 consecutive assessments) or initiation of subsequent therapy (max duration 127.1 weeks).
Population: This analysis was performed in the Safety Analysis Set, which is defined as all patients who received at least 1 or partial dose of melflufen or dexamethasone.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
Participants
  Stringent complete response (sCR) | 0 | 0 | 0
  Complete response (CR) | 0 | 2 | 0
  Very good partial response (VGPR) | 3 | 1 | 0
  Partial response (PR) | 7 | 4 | 1
  Minimal response (MR) | 1 | 1 | 0
  Stable disease (SD) | 5 | 2 | 0
  Progressive disease (PD) | 2 | 0 | 3
  Non-evaluable | 3 | 0 | 0

7. Secondary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is the percentage of patients who achieved a confirmed response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) as best response, as assessed by the Investigator.
Time Frame: Patients were assessed for response after each cycle. After discontinuation of therapy, patients continued to be assessed until disease progression (confirmed on 2 consecutive assessments) (maximum duration 127.1 weeks).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
Participants | 10 | 7 | 1

8. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate (CBR) is the proportion of patients who achieved a confirmed minimal response (MR) or better (stringent complete response [sCR], complete response [CR], very good partial response [VGPR], partial response [PR], and MR) as their best response, as assessed by the Investigator.
Time Frame: Patients were assessed for response after each cycle (maximum duration 127.1 weeks).
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
Participants | 11 | 8 | 1

9. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the date of first study drug (the earliest of melflufen and dexamethasone start date) initiation to the date of first documentation of confirmed PD or death due to any cause, whichever occurred first. Participants were deemed 'progressed' in case of i) unconfirmed progressive disease (PD) as the final response assessment, ii) death after at least one response assessment or PD based on at least two consecutive response assessments at any time, or iii) death before the first response assessment. The distribution of PFS was summarized using the Kaplan-Meier (K-M) method. The median PFS was estimated from the 50th percentile of the corresponding K-M estimates. The 95% confidence interval for median PFS was constructed using the method of Brookmeyer (Brookmeyer, 1982).
Time Frame: Patients were assessed from the initiation of therapy until documented disease progression or initiation of new therapy (maximum duration 127.1 weeks).
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
months | 8.61 [4.30 to 14.52] | 7.66 [6.24 to NA] — Data not estimable. At the final data cut the upper limit CI was not reached at the previous data cut due to too few events | 3.43 [0.95 to NA] — Data not estimable. At the final data cut the upper limit CI was not reached at the previous data cut due to too few events

10. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) is defined as the time from the first evidence of confirmed assessment of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), or partial response (PR) to first confirmed disease progression, or to death due to any cause. The distribution of DOR was summarized using the Kaplan-Meier (K-M) method. The median DOR was estimated from the 50th percentile of the corresponding K-M estimates. The 95% confidence interval for median DOR was constructed using the method of Brookmeyer (Brookmeyer, 1982).
Time Frame: Patients were assessed for response from the first measure of a confirmed response (PR or better) until confirmed progression, death, or initiation of subsequent therapy (maximum duration 127.1 weeks).
Population: This analysis included patients who achieved a best confirmed response of PR or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 10 | 7 | 1
months | 8.31 [5.82 to 23.49] | 13.83 [4.63 to NA] — Data not estimable. At the final data cut the upper limit CI was not reached at the previous data cut due to too few events | NA [NA to NA] — Data not estimable due to an insufficient number of patients. Only one patient had a best response of confirmed PR or better

11. Secondary Outcome: Duration of Clinical Benefit
Description: Duration of clinical benefit (DOCB) was calculated as time in months from the first evidence of confirmed assessment of stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), or minimal response (MR) to first confirmed disease progression, or to death due to any cause. DOCB was defined only for patients with a confirmed MR or better. DOCB was summarized using the Kaplan-Meier (K-M) method. The median DOCB was estimated from the 50th percentile of the corresponding K-M estimates. The 95% confidence interval for median DOCB was constructed using the method of Brookmeyer (Brookmeyer, 1982).
Time Frame: Patients were assessed from the first measure of a confirmed MR or better until confirmed progression, death, or initiation of subsequent therapy (maximum duration 127.1 weeks).
Population: This analysis included patients who achieved a best response of MR or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 11 | 8 | 1
months | 9.26 [5.82 to 23.49] | 10.58 [4.63 to NA] — Data not estimable. At the final data cut the upper limit CI was not reached at the previous data cut due to too few events | NA [NA to NA] — Data not estimable due to an insufficient number of events. Only one patient had a best response of confirmed MR or better.

12. Secondary Outcome: Time to Response
Description: Time from first dose of therapy to first documented confirmed response of partial response (PR) or better.
Time Frame: From initiation of therapy until documented disease response (maximum duration 127.1 weeks).
Population: This analysis included patients who achieved a best confirmed response of PR or better.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 10 | 7 | 1
months | 2.45 [1.0 to 11.3] | 1.18 [0.9 to 7.6] | 2.83 [2.83 to 2.83]

13. Secondary Outcome: Time to Clinical Benefit
Description: Time to clinical benefit was defined as the time from first dose of therapy to first documented confirmed response of minimal response (MR) or better.
Time Frame: as for outcome 6
Population: This analysis included patients who achieved a best response of MR or better.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 11 | 8 | 1
months | 1.12 [1.0 to 8.7] | 1.12 [0.9 to 5.9] | 2.83 [2.83 to 2.83]

14. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from initiation of therapy to death due to any cause. Patients still alive at the end of the study, or lost to follow up, were censored at last day known alive.
Time Frame: Patients were followed for overall survival until death or until the last patient in the study had documented progression (confirmed on 2 consecutive assessments) or initiation of subsequent therapy (maximum of 39.2 months).
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
Number analyzed (Participants) | 21 | 10 | 4
months | 9.76 [5.06 to 15.38] | NA [6.83 to NA] — Data not estimable. Death due to any cause occurred in 3 patients (as reported at both data cuts). The median and upper limit were not reached due to too few events | NA [3.15 to NA] — Data not estimable. Death due to any cause occurred in 1 patient; the patient had a survival time of 3.15 months.The median and upper limit were not reached due to too few events

ADVERSE EVENTS:
Time Frame: SAEs were collected from signing of the ICF until 30 days after the last dose of study treatment or initiation of subsequent therapy, whichever occurred first. Maximum treatment durations for Cohorts 1a, 1b & 2a were 127.1, 94.7 and 36.1 weeks respectively. The AE reporting period is estimated to be 30 days longer.
Description: Non-serious AEs were collected from the start of study treatment until 30 days after the last dose of any study drug or initiation of subsequent therapy, whichever occurred first. The median overall treatment duration for all patients was 25.57 weeks, and the duration of AE reporting is expected to be similar.
Arm/Group | Cohort 1a, Melflufen 40 mg | Cohort 1b, Melflufen 30 mg | Cohort 2a, Melflufen 20 mg
All-Cause Mortality (participants affected / at risk) | 16/21 | 3/10 | 1/4
Serious Adverse Events (participants affected / at risk) | 9/21 | 5/10 | 0/4
Other Adverse Events (participants affected / at risk) | 20/21 | 10/10 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a, Melflufen 40 mg (N=21) | Cohort 1b, Melflufen 30 mg (N=10) | Cohort 2a, Melflufen 20 mg (N=4)
Catheter site haemorrhage (General disorders) | 1 (1) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (8) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Device issue (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1a, Melflufen 40 mg (N=21) | Cohort 1b, Melflufen 30 mg (N=10) | Cohort 2a, Melflufen 20 mg (N=4)
Thrombocytopenia (Blood and lymphatic system disorders) | 14 (79) | 9 (42) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 8 (42) | 5 (17) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (31) | 4 (14) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 2 (5) | 2 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (5) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (6) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (6) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (2) | 4 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0) | 2 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otosalpingitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spondyloarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 3 (8) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Between-group comparisons were not performed in this study due the small number of patients in each cohort, as well as differences with regards to some baseline characteristics.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/10/NCT03639610/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/10/NCT03639610/SAP_001.pdf